CLINICAL TRIAL: NCT05266508
Title: Investigating the Effects of Autonomous Sensory Meridian Response (ASMR) Stimulation on the Functional Connectivity of the Default Mode Network
Brief Title: Effects of ASMR on the Default Mode Network
Status: Completed | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: ASMR-EFF
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Autonomous Sensory Meridian Response; Audiobook
Keywords: Autonomous Sensory Meridian Response; Resting-state fMRI; Default Mode Network

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the effects of Autonomous Sensory Meridian Response (ASMR) stimulation on resting-state brain networks. Therefore, two resting-state fMRI scans are measured in healthy adults. Before each fMRI scan, subjects listen either to ASMR typical sounds or an audio-book (randomized cross-over-design). It is expected to find changes in the functional connectivity of the Default Mode Network caused by passive listening to ASMR.

DETAILED DESCRIPTION:
ASMR describes a phenomenon of a perceived tingling caused by visual or auditory stimulation. This sensation can spread from the neck to the scalp and further to the back and the extremities. The triggering sound often consists of acoustic sounds (crackle, whisper, light nail-tapping) or visual images (e.g., someone is combing their hair), leading to a calm and relaxing feeling. Although ASMR is ubiquitous in platforms like "YouTube", there are just a few studies investigating the effects of ASMR. In one of those studies, Smith and colleagues examined the Default Mode Network of 11 subjects with ASMR stimulation and compared the outcome with a control group consisting of 11 subjects. They found reduced functional connectivity in the ASMR group compared to the control group. Furthermore, the connectivity between the occipital, frontal and temporal cortex was increased.

In the present study, fMRI is used to examine the effects of ASMR stimulation in a randomized cross-over design. Half of the subjects (n=14) receive the ASMR stimulation first, and then the control stimulation (audiobook). The other half of the subjects (n=14) listens to the control stimulation (audiobook) first and afterward to the ASMR stimulation. Typical "tingling" triggering sounds are presented via MRI-compatible headphones. Those sounds can consist of different noises (e.g., whisper, scratching, and knocking).

The primary outcome measure is a change in the functional connectivity of the Default Mode Network as a response to the ASMR stimulation.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 99

Exclusion Criteria:

* mental disorders (dementia, depression)
* MRI contraindications
* claustrophobia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects aged 18 to 99
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Changed functional connectivity | 45 minutes
  Functional connectivity is measured using resting-state fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Jens D. Rollnik, MD, Study Director — BDH-Clinik Hessisch Oldendorf
Locations (1):
- BDH-Clinic Hessisch Oldendorf, Hessisch Oldendorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith SD, Fredborg BK, Kornelsen J. Atypical Functional Connectivity Associated with Autonomous Sensory Meridian Response: An Examination of Five Resting-State Networks. Brain Connect. 2019 Jul;9(6):508-518. doi: 10.1089/brain.2018.0618. Epub 2019 May 7. PMID 30931592